CLINICAL TRIAL: NCT01382914
Title: Determination of a Threshold for Mouth Rinse Induced Discoloration of Teeth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: PAR01-2011
Record Dates: First submitted 2011-06-24; First posted 2011-06-27 (Estimated); Last update posted 2012-01-18 (Estimated); Status verified 2012-01

CONDITIONS: Discoloration of Teeth
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chlorhexidine 0.12 % (Experimental)
  Interventions: Other: chlorhexidine 0.12%

INTERVENTIONS:
Other: chlorhexidine 0.12% — twice daily, 10 ml, topical
  Other Names: Perio-Aid 0.12%

SUMMARY:
The purpose of this study is to daily monitor the discoloration of teeth when participants rinse with a mouth rinse and black tea and to determine the time point when unacceptable discoloration occurs.

DETAILED DESCRIPTION:
Tooth discoloration is a side effect of most mouth rinse solutions. It impairs the aesthetic appearance especially of the front teeth. The aim of this pilot study is to determine a time point when visible discoloration appears in the front teeth. Therefore, participants of this study will rinse twice daily with chlorhexidine mouth rinse for 10 days. To elicit a more pronounced discoloration, participants will rinse with black tea right after the chlorhexidine rinse. Discoloration will be measured daily by discoloration index, by spectrophotometry, and by the use of a digital photo.

ELIGIBILITY:
Inclusion Criteria:

* persons aged 18 to 30 years
* written informed consent
* healthy participants
* participants who have no or mild gingivitis
* participants who have all incisors and canines in the upper and lower jaw

Exclusion Criteria:

* participants who have severe general diseases
* participants who have allergies against the ingredients of the mouthrinse
* participants who are enrolled in another clinical study
* participants who are not able to oversee the consequences of the study
* female participants who are pregnant or breast feeding
* participants who have impaired compliance
* participants who have moderate or severe gingivitis
* participants who have fillings in the incisors and canines
* participants who smoke

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Time point (day) when delta E > 2 | 11 days

SECONDARY OUTCOMES:
Time point (day) when discoloration index changes compared to baseline | 11 days
Time point (day) when changes in the photo evaluation occur compared to baseline | 11 days
Time point (day) when discoloration occurs subjectively (questionnaire) compared to baseline | 11 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hoffmann, Prof. Dr., Principal Investigator — Technische Universität Dresden
Locations (1):
- Dreden University of Technology, Universitätsklinikum, Poliklinik für Parodontologie, Dresden, Saxony, Germany

REFERENCES:
- [Background] Addy M, Prayitno S, Taylor L, Cadogan S. An in vitro study of the role of dietary factors in the aetiology of tooth staining associated with the use of chlorhexidine. J Periodontal Res. 1979 Sep;14(5):403-10. doi: 10.1111/j.1600-0765.1979.tb00238.x. No abstract available. PMID 161782
- [Background] Bengel WM. Digital photography and the assessment of therapeutic results after bleaching procedures. J Esthet Restor Dent. 2003;15 Suppl 1:S21-32; discussion S32. doi: 10.1111/j.1708-8240.2003.tb00315.x. PMID 15000901
- [Background] Denissen H, Dozic A. Photometric assessment of tooth color using commonly available software. Eur J Esthet Dent. 2010 Summer;5(2):204-15. PMID 20589263